CLINICAL TRIAL: NCT00800826
Title: The Combination Effect of Dexmedetomidine and Morphine in Postoperative Patient-Controlled Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 950910
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2008-12

CONDITIONS: Analgesia, Patient-Controlled; Analgesia, Postoperative
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: dexmedetomidine

SUMMARY:
This study was designed to examine the analgesic and side effects of dexmedetomidine-morphine mixture for intravenous patient-controlled analgesia (PCA).

DETAILED DESCRIPTION:
Patient-controlled analgesia (PCA) is a widely accepted method to control postoperative pain. Morphine is the commonest opioid for PCA, however its side effects are troublesome. Morphine-related side effects include pruritus, nausea, vomiting, constipation, urinary retention, respiratory depression, and sedation. Many studies had been conducted to reduce the side effect of morphine. The current trend of reducing morphine side effect is direct combination of other drugs and morphine in PCA. The advantages of this method are convenient in clinical use and preventive for side effects. Dexmedetomidine is a highly selec¬tive α2-adrenergic receptor agonist that has been reported to cause sedative effects and reduce opioid requirements in the perioperative period. The main advantage of this drug is that it does not cause serious respiratory side effects. The analgesic, sedative/hypnotic and anxiolytic prop¬erties of dexmedetomidine make this drug potentially useful for postoperative sedation and analgesia. No previous study had investigated the effect of direct combination of dexmedetomidine and morphine in PCA. The goal of this study is to investigate the combination effect of dexmedetomidine and morphine in postoperative patient-controlled analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign informed consent to receive general anesthesia and postoperative analgesia with a PCA device
2. Age between 18-65 y/o
3. ASA physical status I-III
4. Scheduled surgical procedures: gynecological surgery (vaginal or abdominal total hysterectomy), general surgery (gastrectomy, hepatectomy, colon cancer) , orthopedic (spinal fusion or total knee placement), or neurosurgical (cervical decompression)

Exclusion Criteria:

1. Patients with a definite diagnosis of chronic pain syndrome, psychiatric disorders, or drug abuse (include opioids, NSAIDs, sedatives, antidepressants).
2. Use of sedatives, analgesics, antiemetics, or antipruritics within 24 hours before operation.
3. Patients with definite diagnosis of esophageal reflux syndrome.
4. Patients with the probability to be pregnant.
5. Intraoperative fentanyl use > 6 μg/kg.
6. Patients with significant bradycardia (HR < 60/min) and hypotension (SBP < 90mmHg) after the surgery.
7. The duration of surgery is longer than 6 hours.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-11; Study Completion 2008-04 (Actual)